CLINICAL TRIAL: NCT04188041
Title: Improving Rhode Island's Tuberculosis Preventive Services in Primary Care: A Mixed-Methods Evaluation of an Innovative Telementoring Model
Brief Title: Improving Rhode Island's Tuberculosis Preventive Services in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent Hospital, Rhode Island (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Daria Szkwarko, Assistant Professor, Family Medicine, Kent Hospital, Rhode Island
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 1370981-4; U54GM115677 (NIH)
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-06

CONDITIONS: Latent Tuberculosis
Keywords: Project ECHO; primary care
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: 25 primary care team members will be purposively sampled to undergo key informant interviews regarding LTBI testing and treatment knowledge, attitudinal, and skill gaps. Then, 12 primary care team members will be recruited to participate in a virtual six-month TB infection ECHO course. Participants will be asked to complete quantitative surveys before and after the course as well as post-session surveys following each session. Paired data from pre- and post-course surveys will be analyzed accordingly depending on the distribution of results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qualitative (No Intervention): Specific Aim 1: Explore the specific knowledge, attitudinal, and skills gaps to TB infection testing and treatment among primary care team members in RI through qualitative key informant interviews.
  In Aim 1, 25 primary care team members from the Brown Family Medicine and Care New England networks will be purposively sampled to undergo key informant interviews regarding TB infection testing and treatment knowledge, attitudinal, and skill gaps. Questions will be asked to ascertain gaps throughout the entire latent TB infection care cascade. The results from Aim 1 will be used to design the survey instrument and the curriculum for an innovative, telementoring program (TB infection ECHO).
- Quantitative (Other): Specific Aim 2: Design and evaluate an evidence-based telementoring intervention (ECHO model) that addresses the identified TB infection gaps in Aim 1, and evaluate this model for feasibility as well as its impact on primary care team member knowledge and TB infection testing and treatment in RI. 12 primary care team members will be recruited to participate in a virtual six-month TB infection ECHO course. Participants will be asked to complete quantitative surveys before and after the course as well as post-session surveys following each session. Survey questions will assess feasibility measures related to process, resources, and management and impact measures related to learning and performance. Paired data from pre- and post-course surveys will be analyzed accordingly depending on the distribution of results.
  Interventions: Other: TB Infection ECHO
- Retrospective chart review (Other): Pilot a retrospective electronic medical record (EMR) data review to examine RI primary care providers' testing and treatment before and after ECHO implementation and evaluate the model's reach. In Aim 3, data will be retrospectively extracted from two participants' clinics to research RI primary care providers' testing and treatment patterns before and after the ECHO course. The two clinics will be identified once Aim 2 is completed.
  Interventions: Other: TB Infection ECHO

INTERVENTIONS:
Other: TB Infection ECHO — A six-month virtual telementoring course regarding TB infection testing and treatment that incorporates didactics, case presentation, and discussion
  Arms: Quantitative; Retrospective chart review

SUMMARY:
This study explores primary care team members' knowledge, attitudinal, and skill gaps related to latent tuberculosis infection (LTBI) testing and treatment. The gaps identified will inform the design of a survey and telementoring educational program (tuberculosis (TB) infection ECHO course). The EMR data query will further explore the reach of the expansion for community healthcare outcomes (ECHO) model. The hypothesis for this study is that the TB infection ECHO course will be feasible, will have a significant impact on primary care provider participants' learning and performance related to LTBI testing and treatment in their primary care practices, and will increase the number of LTBI tests and treatment prescribed in primary care.

DETAILED DESCRIPTION:
This pilot study will use a mixed-methods design called an exploratory sequential translational research design. In this type of study design, the initial qualitative phase informs the design of an intervention (in this case a TB infection ECHO) and an instrument (in this case structured surveys) to study the intervention. The third phase implements the designed intervention and/or instrument to collect data and quantitatively assess the outcomes of interest (in this case feasibility and impact). The final aspect of the third phase explores an EMR data query to assess the reach of the intervention (providers' testing and treatment in the real world). In Aim 1, 25 primary care team members from our Brown Family Medicine, Care New England, and federally qualified health center networks will be purposively sampled to undergo key informant interviews regarding LTBI testing and treatment knowledge, attitudinal, and skill gaps. Questions will be asked to ascertain gaps throughout the entire latent TB infection care cascade. The results from Aim 1 will be used to design the survey instrument and the curriculum for an innovative, telementoring program (TB infection ECHO). In Aim 2, 12 primary care team members will be recruited to participate in a virtual six-month TB infection ECHO course. Participants will be asked to complete quantitative surveys before and after the course as well as post-session surveys following each session. Survey questions will assess feasibility measures related to process, resources, and management and impact measures related to learning and performance. Paired data from pre- and post-course surveys will be analyzed accordingly depending on the distribution of results. In Aim 3, data will be extracted from two ECHO participants' clinic sites before, during, and after ECHO implementation. Data will include information about LTBI testing and treatment to understand the reach and impact of the intervention of providers' testing and treatment behavior. This study will lead to an ECHO research framework that can be used for future ECHO courses that address other diseases in Rhode Island (RI).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Primary care team members in Rhode Island including doctors, nurses, nurse practitioners, physician assistants, or other healthcare providers who are involved in primary care.

Exclusion Criteria:

* < 18 years of age
* Primary care team members who do not primarily work in Rhode Island

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown Family Medicine Department, Pawtucket, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Aim 1: one participant was excluded because it turned out they did not actually conduct primary care which was an inclusion criterion.
  Aim 2: completing the pre and post surveys was voluntary after consent. Several participants did not voluntarily complete both surveys.
  Aim 3: retrospective chart review was only completed for one site before the ECHO course
Groups:
- Aim 1: Key Informant Interviews: Primary care team members who consented to participate in key informant interviews regarding their knowledge, attitudes, and skills about latent tuberculosis infection testing and treatment.
- Aim 2: RI LTBI ECHO Participants: Rhode Island (RI) Primary care team members who participated in the Rhode Island Latent Tuberculosis ECHO program and consented to be part of aim 2. Participants were asked to complete a pre and post course survey.
- Aim 3: Retrospective Chart Review: A retrospective chart review was completed at Blackstone Valley Community Health Center to review LTBI treatment patterns among primary care providers. An EMR query was performed for patients > 18 years who had a documented interferon gamma release assay test or TST and/or ICD-10 codes for LTBI between April 2019 and April 2020.
Period: Aim 1: Key Informant Interviews
Arm/Group | Aim 1: Key Informant Interviews | Aim 2: RI LTBI ECHO Participants | Aim 3: Retrospective Chart Review
Started | 25 | 0 | 0
Completed | 24 | 0 | 0
Not Completed | 1 | 0 | 0
Period: Aim 2: RI LTBI ECHO Program Participants
Arm/Group | Aim 1: Key Informant Interviews | Aim 2: RI LTBI ECHO Participants | Aim 3: Retrospective Chart Review
Started | 4 | 8 | 0
Completed | 3 | 5 | 0
Not Completed | 1 | 3 | 0
Period: Aim 3: Retrospective Chart Review
Arm/Group | Aim 1: Key Informant Interviews | Aim 2: RI LTBI ECHO Participants | Aim 3: Retrospective Chart Review
Started | 0 | 0 | 51
Completed | 0 | 0 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Aim 3 (retrospective chart review) data were collected from an electronic medical record (EMR) and were de-identified in nature.
  Credentials were not collected so cannot be provided.
Groups:
- Aim 1: Key Informant Interviews: RI Primary care team members who consented to participate in key informant interviews regarding their knowledge, attitudes, and skills about latent tuberculosis infection testing and treatment.
- Aim 2: RI LTBI ECHO Participants: Some as well as several new individuals participated in the Rhode Island Latent Tuberculosis ECHO program and consented to be part of aim 2. Participants were asked to complete a pre and post course survey.
- Aim 3: Retrospective Chart Review: Individuals > 18 years identified via a retrospective chart review who had a positive interferon gamma release assay test or TST and/or ICD-10 codes for LTBI between April 2019 and April 2020.
- Total: Total of all reporting groups
Arm/Group | Aim 1: Key Informant Interviews | Aim 2: RI LTBI ECHO Participants | Aim 3: Retrospective Chart Review | Total
Number analyzed (Participants) | 25 | 8 | 51 | 84
Age, Categorical [Count of Participants; unit: Participants] — Population: one participant's age is unknown
  Participants
    Aim 1: number analyzed (Participants) | 21 | 4 | 0 | 25
    Aim 1: <=18 years | 0 | 0 | 0 | 0
    Aim 1: Between 18 and 65 years | 21 | 3 | 0 | 24
    Aim 1: >=65 years | 0 | 1 | 0 | 1
    Aim 2: number analyzed (Participants) | 0 | 7 | 0 | 7
    Aim 2: <=18 years | 0 | 0 | 0 | 0
    Aim 2: Between 18 and 65 years | 0 | 7 | 0 | 7
    Aim 2: >=65 years | 0 | 0 | 0 | 0
    Aim 3: number analyzed (Participants) | 0 | 0 | 51 | 51
    Aim 3: <=18 years |  |  | 0 | 0
    Aim 3: Between 18 and 65 years |  |  | 43 | 43
    Aim 3: >=65 years |  |  | 8 | 8
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 4 individuals from Aim 1 also participated in Aim 2. 8 individuals only participated in Aim 2.
  Participants
    Aim 1: Key Informant Interviews: number analyzed (Participants) | 21 | 4 | 0 | 25
    Aim 1: Key Informant Interviews: Female | 12 | 2 | 0 | 14
    Aim 1: Key Informant Interviews: Male | 9 | 2 | 0 | 11
    Aim 2: RI LTBI ECHO Participants: number analyzed (Participants) | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: Female | 0 | 5 | 0 | 5
    Aim 2: RI LTBI ECHO Participants: Male | 0 | 3 | 0 | 3
    Aim 3: Retrospective Chart Review: number analyzed (Participants) | 0 | 0 | 51 | 51
    Aim 3: Retrospective Chart Review: Female | 0 | 0 | 37 | 37
    Aim 3: Retrospective Chart Review: Male | 0 | 0 | 14 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 4 individuals from Aim 1 also participated in Aim 2. 8 individuals only participated in Aim 2.
  Participants
    Aim 1: Key Informant Interviews: number analyzed (Participants) | 21 | 4 | 0 | 25
    Aim 1: Key Informant Interviews: Hispanic or Latino | 2 | 0 | 0 | 2
    Aim 1: Key Informant Interviews: Not Hispanic or Latino | 19 | 4 | 0 | 23
    Aim 1: Key Informant Interviews: Unknown or Not Reported | 0 | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: number analyzed (Participants) | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: Hispanic or Latino | 0 | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: Not Hispanic or Latino | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: Unknown or Not Reported | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: number analyzed (Participants) | 0 | 0 | 51 | 51
    Aim 3: Retrospective Chart Review: Hispanic or Latino | 0 | 0 | 24 | 24
    Aim 3: Retrospective Chart Review: Not Hispanic or Latino | 0 | 0 | 27 | 27
    Aim 3: Retrospective Chart Review: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 4 individuals from Aim 1 also participated in Aim 2. 8 individuals only participated in Aim 2.
  Participants
    Aim 1: Key Informant Interviews: number analyzed (Participants) | 21 | 4 | 0 | 25
    Aim 1: Key Informant Interviews: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Aim 1: Key Informant Interviews: Asian | 2 | 0 | 0 | 2
    Aim 1: Key Informant Interviews: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Aim 1: Key Informant Interviews: Black or African American | 0 | 0 | 0 | 0
    Aim 1: Key Informant Interviews: White | 18 | 4 | 0 | 22
    Aim 1: Key Informant Interviews: More than one race | 1 | 0 | 0 | 1
    Aim 1: Key Informant Interviews: Unknown or Not Reported | 0 | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: number analyzed (Participants) | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: American Indian or Alaska Native |  | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: Asian |  | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: Black or African American |  | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: White |  | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: More than one race |  | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: Unknown or Not Reported |  | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: number analyzed (Participants) | 0 | 0 | 51 | 51
    Aim 3: Retrospective Chart Review: American Indian or Alaska Native |  |  | 0 | 0
    Aim 3: Retrospective Chart Review: Asian |  |  | 1 | 1
    Aim 3: Retrospective Chart Review: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
    Aim 3: Retrospective Chart Review: Black or African American |  |  | 17 | 17
    Aim 3: Retrospective Chart Review: White |  |  | 4 | 4
    Aim 3: Retrospective Chart Review: More than one race |  |  | 1 | 1
    Aim 3: Retrospective Chart Review: Unknown or Not Reported |  |  | 28 | 28
Region of Enrollment [Number; unit: participants]
  United States | 25 | 8 | 51 | 33
Years out of training [Count of Participants; unit: Participants] — Population: 4 individuals from Aim 1 also participated in Aim 2. 8 individuals only participated in Aim 2.
  Participants
    Aim 1: Key Informant Interviews: number analyzed (Participants) | 21 | 4 | 0 | 25
    Aim 1: Key Informant Interviews: In training | 3 | 0 | 0 | 3
    Aim 1: Key Informant Interviews: < 5 years out of training | 12 | 1 | 0 | 13
    Aim 1: Key Informant Interviews: 5 or more years out of training | 3 | 3 | 0 | 6
    Aim 1: Key Informant Interviews: unknown | 3 | 0 | 0 | 3
    Aim 2: RI LTBI ECHO Participants: number analyzed (Participants) | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: In training | 0 | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: < 5 years out of training | 0 | 3 | 0 | 3
    Aim 2: RI LTBI ECHO Participants: 5 or more years out of training | 0 | 3 | 0 | 3
    Aim 2: RI LTBI ECHO Participants: unknown | 0 | 2 | 0 | 2
    Aim 3: Retrospective Chart Review: number analyzed (Participants) | 0 | 0 | 51 | 51
    Aim 3: Retrospective Chart Review: In training | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: < 5 years out of training | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: 5 or more years out of training | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: unknown | 0 | 0 | 51 | 51
Credentials [Count of Participants; unit: Participants] — Credentials of the participant to distinguish whether they are a primary care clinician (MD, DO, NP) vs a nurse (RN). Population: 4 individuals from Aim 1 also participated in Aim 2. 8 individuals only participated in Aim 2.
  Participants
    Aim 1: Key Informant Interviews: number analyzed (Participants) | 21 | 4 | 0 | 25
    Aim 1: Key Informant Interviews: Primary care clinician | 18 | 4 | 0 | 22
    Aim 1: Key Informant Interviews: Nurse | 3 | 0 | 0 | 3
    Aim 1: Key Informant Interviews: Not Applicable | 0 | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: number analyzed (Participants) | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: Primary care clinician | 0 | 8 | 0 | 8
    Aim 2: RI LTBI ECHO Participants: Nurse | 0 | 0 | 0 | 0
    Aim 2: RI LTBI ECHO Participants: Not Applicable | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: number analyzed (Participants) | 0 | 0 | 51 | 51
    Aim 3: Retrospective Chart Review: Primary care clinician | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: Nurse | 0 | 0 | 0 | 0
    Aim 3: Retrospective Chart Review: Not Applicable | 0 | 0 | 51 | 51

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Participant Attendance
Description: Number of consented participants attending each expansion for community healthcare outcomes (ECHO) session who consented to participate in the course
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: The number of consented participants who attended the RI LTBI ECHO program
Measure: Number; unit: participants
Groups:
- RI LTBI ECHO Program Participants: RI Primary care team members who participated in the Rhode Island Latent Tuberculosis ECHO program and consented to be part of aim 2. Participants were asked to complete a pre and post course survey.
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 12
participants
  Launch Session | 10
  Session 1 | 9
  Session 2 | 7
  Session 3 | 8
  Session 4 | 8
  Session 5 | 8
  Session 6 | 6

2. Primary Outcome: Feasibility: Participant Retention
Description: Percentage of registered participants attending one of the last two ECHO sessions
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Number of consented participants who attended sessions 5 or 6
Measure: Count of Participants; unit: Participants
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 12
Participants | 9

3. Primary Outcome: Impact: Procedural Knowledge
Description: Change in participants' confidence in assessing a patient's risk for tuberculosis (TB) infection based on a likert scale rating (1=not at all confident and 5=extremely confident) included in the pre- and post- structured surveys administered before and after the ECHO intervention.
Time Frame: Pre-survey was emailed 2 weeks prior to the course and could be filled out anytime before a participant attended their first session. The post-survey was emailed immediately following the final session (3/4/2021) and were completed within three weeks.
Population: Consented Survey Participants who participated in the RI LTBI ECHO and responded to the pre-survey and/or post-survey question. "Please rate your confidence in performing each of the areas of latent TB infection practice below: Assessing a patient's risk for TB infection" 1=Not at all confident, 2=Not very confident, 3=moderately confident, 4=very confident, 5=extremely confident
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 12
score on a scale
  Pre-Survey | 3.09 (0.51)
  Post-Survey | 4.25 (0.66)
Statistical Analysis 1: Comparison: RI LTBI ECHO Program Participants; Non-parametric Wilcoxon signed rank test for paired data was used to test for significant change in confidence; Test type: Other — see above; p = 0.02, Wilcoxon signed rank test

4. Primary Outcome: Impact: Self-reported LTBI Screening Percentage by Participants on Pre- and Post-ECHO Course Surveys
Description: Change in participants' self-reported estimates of patients screened for TB infection. Participants estimated their screening percentage on a sliding scale from 0-100%. Mean estimates will be calculated for the pre- and post- structured survey responses administered before and after the ECHO intervention.
Time Frame: as for outcome 3
Population: Consented participants who responded to both pre- and post-surveys were asked to participate voluntarily. All 12 participants answered some of the pre-survey questions (only 6 answered the question of interest). Out of the 12, only 8 responded to the post survey. Of the 8, 7 answered the question of interest.
Measure: Mean (Standard Deviation); unit: percentage of patients screened
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 12
percentage of patients screened
  Pre-Survey: number analyzed (Participants) | 6
  Pre-Survey | 45.67 (38.6)
  Post Survey: number analyzed (Participants) | 7
  Post Survey | 25.86 (25.99)

5. Primary Outcome: Impact: Participants' Self-reported LTBI Treatment Percentages on Pre- and Post ECHO Surveys
Description: Change in participants' self-reported estimates of patients treated for TB infection. Participants will estimate the percentage of patients started on any TB treatment on a sliding scale from 0-100%. Mean percentages will be calculated between the pre- and post- structured survey responses administered before and after the ECHO intervention.
Time Frame: Pre-survey was emailed two weeks prior to the course and could be filled out anytime before a participant attended their first session. The post-survey was emailed immediately following the final session on 3/4/2021 and were completed within three weeks.
Population: Participation in the surveys was voluntary so not all participants answered all questions. All 12 participants answered some of the pre-survey questions (only 4 answered the question of interest). Out of the 12, only 8 responded to the post survey. Of those 8, 5 answered the question of interest.
Measure: Mean (Standard Deviation); unit: percentage of patients started on tx
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 12
percentage of patients started on tx
  Pre-Survey: number analyzed (Participants) | 4
  Pre-Survey | 50 (50)
  Post-Survey: number analyzed (Participants) | 5
  Post-Survey | 11 (19.6)

6. Primary Outcome: Reach: LTBI Testing
Description: Proportion(# of TB tests/# of visits) of patients tested for LTBI in a health center population before, during and after ECHO implementation to assess providers' behavior change. This data will be obtained from an electronic medical record data query
Time Frame: Three-months prior, ECHO course, three- months post
Population: data were not collected
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 0

7. Primary Outcome: Reach: LTBI Treatment
Description: Patient level LTBI treatment before, during and after ECHO implementation to assess providers' behavior change. Proportion(# of TB treatment initiated/# of patients diagnosed with LTBI) of patients treated for LTBI in a health center population before, during and after ECHO implementation to assess providers' behavior change. This data will be obtained from an electronic medical record data query.
Time Frame: Three-months prior, ECHO course, three- months post
Population: data were not collected
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Feasibility: Case Submission
Description: Percentage of cases submitted by participants on time during the ECHO course
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Participants who were asked to submit a case
Measure: Count of Participants; unit: Participants
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 6
Participants | 6

9. Secondary Outcome: Feasibility: ECHO Session Timing
Description: Percentage of participants' who agree that session timing was convenient. This will be collected monthly from post-session surveys via a likert scale (1=strongly disagree and 5=strongly agree)
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Data were not collected
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Feasibility: Connectivity
Description: Percentage of participants' who agree that connectivity was adequate during the ECHO session. This will be collected monthly from post-session surveys via a likert scale (1=strongly disagree and 5=strongly agree)
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Data were not collected
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Feasibility: Videoconferencing Equipment
Description: Percentage of participants' who agree that videoconferencing equipment was adequate during the ECHO session. This will be collected monthly from post-session surveys via a likert scale (1=strongly disagree and 5=strongly agree)
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Data were not collected
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Feasibility: Content Expert Facilitation
Description: Participants rating of whether the speaker demonstrated excellent educational skills. This will be collected monthly from post-session surveys via a likert scale (1=strongly disagree and 5=strongly agree)
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Participation in post session evaluations was voluntary. Not all 9 consented participants who completed any of the evaluations completed all of the evaluations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- RI LTBI ECHO Program Participants: RI Primary care team members who participated in the Rhode Island Latent Tuberculosis ECHO program and consented to be part of aim 2. Participants were asked to complete post session evaluations.
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 9
score on a scale
  Session 1: number analyzed (Participants) | 6
  Session 1 | 4.83 (0.41)
  Session 2: number analyzed (Participants) | 7
  Session 2 | 4.86 (0.38)
  Session 3: number analyzed (Participants) | 7
  Session 3 | 4.43 (0.79)
  Session 4: number analyzed (Participants) | 7
  Session 4 | 4.71 (0.49)
  Session 5: number analyzed (Participants) | 6
  Session 5 | 4.83 (0.41)
  Session 6: number analyzed (Participants) | 6
  Session 6 | 4.33 (0.82)

13. Secondary Outcome: Feasibility: Communication With ECHO Hub
Description: Percentage of participants' who agree that the communication with the ECHO hub team was adequate during the ECHO session. This will be collected monthly from post-session surveys via a likert scale (1=strongly disagree and 5=strongly agree)
Time Frame: Session 1 10/8/20; Session 2 11/5/20; Session 3 12/10/20; Session 4 1/7/21; Session 5 2/4/21; Session 6 3/4/21
Population: Data were not collected
Arm/Group | RI LTBI ECHO Program Participants
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Primary Care Providers' and Nurses' Reported Frequency in Conducting LTBI Screening
Description: Qualitative interviews were conducted with primary care providers and nurses in RI regarding their knowledge, attitudes, and skills regarding LTBI management. A key focus of the interview was related to frequency of conducting LTBI screening. Here we summarize the frequency of providers and nurses who reported never conducting TB screening, infrequently conducting TB screening, or frequently conducting TB screening.
Time Frame: Interviews were conducted between October 2, 2019 and June 17, 2020
Measure: Count of Participants; unit: Participants
Groups:
- Aim 1: Key Informant Interviewees: Primary care team members who consented to participate in key informant interviews regarding their knowledge, attitudes, and skills about latent tuberculosis infection testing and treatment
Arm/Group | Aim 1: Key Informant Interviewees
Number analyzed (Participants) | 24
Participants
  Never conduct TB screening | 3
  Infrequently conduct TB screening | 14
  Frequently conduct TB screening | 7

ADVERSE EVENTS:
Description: Adverse events were not collected since the intervention in this study was educational in nature.
Arm/Group | RI LTBI ECHO Program Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT04188041/Prot_SAP_000.pdf